CLINICAL TRIAL: NCT04357171
Title: Multi-center, Randomized, Parallel-group, Superiority Study to Compare Outcomes of Protective Double-Barrelled Colostomy Versus Protective Double-Barrelled Ileostomy in Low Anterior Resection for Rectal Cancer
Brief Title: PReventive cOlostomy vs Ileostomy in Low anTErior reCTal Resection
Acronym: PROTECT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Russian Society of Colorectal Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 5
Record Dates: First submitted 2020-04-20; First posted 2020-04-22 (Actual); Last update posted 2020-04-22 (Actual); Status verified 2020-04

CONDITIONS: Rectal Cancer
Keywords: colostomy; ileostomy; rectal cancer; low anterior resection
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ileostomy (Active Comparator): Loop protective ileostomy as a defunction mean after low anterior resection with D3 lymphnode dissection
  Interventions: Procedure: Low anterior resection with protective loop ileostomy
- Colostomy (Active Comparator): Loop protective transverse colostomy as a defunction mean after low anterior resection with D3 lymphnode dissection
  Interventions: Procedure: Low anterior resection with protective loop transverse colostomy

INTERVENTIONS:
Procedure: Low anterior resection with protective loop ileostomy — Nerve-sparing paraaortic lymph node dissection is performed. The inferior mesenteric artery is divided at 1-2 cm from its origin from the aorta or right below left colic artery. Nerve-sparing total mesorectal excision is performed. Side-to-end sigmoido-rectal anastomosis is created. A loop defunctioning ileostomy is performed.
  Arms: Ileostomy
Procedure: Low anterior resection with protective loop transverse colostomy — Nerve-sparing paraaortic lymph node dissection is performed. The inferior mesenteric artery is divided at 1-2 cm from its origin from the aorta or right below left colic artery. Nerve-sparing total mesorectal excision is performed. Side-to-end sigmoido-rectal anastomosis is created. A loop defunctioning transverse colostomy is performed.
  Arms: Colostomy

SUMMARY:
The type of preventive intestinal stoma (colostomy/ileostomy) after low anterior rectal resection rectum is still a debate.

This study purpose is to demonstrate that preventive loop ileostomy is characterized by a higher readmission rate caused by dehydration, in comparison with the loop colostomy.

DETAILED DESCRIPTION:
Modern surgery for the rectal cancer is featured by sphincter-preserving operations. It is proved that colorectal anastomosis leakage is severe and, in some cases, lethal complication that reduces quality of life of patients and increases the risk of disease reccurence.

The presence of preventive stoma is an effective way to avoid this complication that is why it's included to treatment protocols for the middle and low ampullary rectal cancers is undisputed by the most of surgeons. However, the type of preventive stoma is under discussion yet and remains to be an urgent issue.

The majority of large meta-analyzes demonstrates that preventive ileostomy is used more often for the protection of low colorectal anastomoses. In the western countries the preferred method is double barreled ileostomy due to more rapid formation and closure, as well as due to lower rate of stoma-related morbidity.

In Russia and CIS countries the double-barreled transverse colostomy is a preferred method of defuction of low colorectal anastomosis due to lower rate of electrolytic disorders and related hospital admissions, along with series of unproven advantages.

Presented study will allow to reveal the early and late postoperative morbidity rate and the related hospital re-admissions in real-life clinical practice of Russia from the standpoints of evidence- based medicine, to define indications and contraindications for each type of "low" colorectal anastomosis protection with the least risk for the patient.

ELIGIBILITY:
Inclusion Criteria:

* Mid- and low rectal cancer
* Age ≧ 18
* TME
* ASA ≦ 3
* No previous stoma formation
* Informed consent for participation

Exclusion Criteria:

* Patients lost during the follow-up
* Refusal of the patient from further participation in the study
* Inability of stoma formation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2012-01-14 (Actual); Primary Completion 2020-02-02 (Actual); Study Completion 2020-02-02 (Actual)

PRIMARY OUTCOMES:
The rate of readmissions due to severe dehydratation | 6 weeks
  The percentage of patients who were readmitted to the hospital due to dehydration, that could not be managed in outhospital setting

SECONDARY OUTCOMES:
Early postoperative complications rate | 30 days after the initial procedure
  The rate of all postoperative complications in early postoperative period after resectional surgery
Late postoperative complications rate | starting on 31st day and within 6 months in late postoperative period after the initial procedure
  The rate of all postoperative complications
Overall quality of life | 6 and 12 months after the initial procedure
  Assessed with patient-reported questionnaire SF-36. A total score in each of 8 sections will be calculated and transformed into a 0-100 scale with a score of zero equivalent to maximum disability and a score of 100 equivalent to no disability
Time with stoma | 5 years
  The period of time between initial resectional procedure and closure of protetctive stoma only in patients who had their intestinal stoma reversed
The rate of early postoperative complications after stoma closure operation | 3 months after stoma closure
  The rate of early postoperative complications after stoma closure operation

CONTACTS AND LOCATIONS:
Overall Officials: Petr Tsarkov, Principal Investigator — Clinic of Colorectal and Minimally Invasive Surgery; Inna Tulina, Study Chair — Clinic of Colorectal and Minimally Invasive Surgery